CLINICAL TRIAL: NCT03183102
Title: The Role of the Gut Microbiota in Estrogen Metabolism and Dietary Flax as a Potential Modulator.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 16-6978H
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Menopause
MeSH Terms: interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Biological samples will be masked for endpoint analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Estrogen suppression no flax (No Intervention): Control subjects will not consume flaxseed, but will receive GnRH suppression
- Estrogen suppression with flax (Experimental): Flax subjects will consume flaxseed for 2 months in addition to GnRH suppression
  Interventions: Dietary Supplement: Flaxseed

INTERVENTIONS:
Dietary Supplement: Flaxseed — 2 months of dietary flaxseed supplementation
  Arms: Estrogen suppression with flax

SUMMARY:
The purpose of this pilot study is to determine if suppressing estrogen in premenopausal women results in changes in gut microbiota and if dietary flaxseed modulates these changes.

DETAILED DESCRIPTION:
This pilot study will begin to address whether gut microbiota change with estrogen suppression. Specifically, the investigators will test whether gut microbial diversity and abundance change in response to estrogen suppression and consumption of dietary flaxseed. To test this possibility the investigators will recruit premenopausal women (age 20-40 years old)and collect fecal samples before and after 1 month of estrogen suppression with GnRH agonist. The investigators will analyze the gut microbiota in response to estrogen loss and whether this differs with the consumption of flaxseed.

ELIGIBILITY:
Inclusion Criteria:

* healthy premenopausal women (20-40 years)
* normal to overweight (22-29.9 kg/m2)
* normally menstruating (25-35 day cycles)
* not have used estrogen-based contraception for >6 months.
* sedentary to moderately active (exercise ≤120 min week-1)
* must not be taking phytoestrogenic dietary supplements, or lipid- or glucose- lowering medications.

Exclusion Criteria:

* smoking
* pregnancy or breastfeeding
* Hormonal contraceptive use (past 6 mo.)
* Women with contraindications to GnRHAG:
* History of fragility fracture
* Low BMD (i.e., proximal femur or lumbar spine z scores < -2.0)
* Abnormal vaginal bleeding
* History of breast cancer or other estrogen-dependent neoplasms
* History of venous thromboembolic events
* Hypersensitivity to leuprolide acetate or benzyl alcohol (the vehicle for injection of leuprolide acetate)
* Evidence for depressive symptoms (Score ≥ 18 on the Beck Depression Inventory, BDI)
* Moderate or severe renal impairment defined as a calculated creatinine clearance <50 mL/min based on the equation of Cockcroft and Gault91
* Chronic hepatobiliary disease, conservatively defined as liver function tests (AST, ALT, alkaline phosphatase, Total Bilirubin) >1.5 times the upper limit of normal (if such values are obtained on initial screening and thought to be transient in nature, repeated testing will be allowed)
* antibiotic or probiotic use within 2 months of sample collection

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change in gut microbiota diversity | At baseline (day 0) and 30 days after estrogen suppression, with and without dietary flaxseed 30 days before estrogen suppression and during the 30 days of estrogen suppression
  16s rRNA sequencing--Illumina MiSeq

SECONDARY OUTCOMES:
Estrogen metabolites | At baseline (day 0) and 30 days after estrogen suppression, with and without dietary flaxseed 30 days before estrogen suppression and during the 30 days of estrogen suppression
  estrogen metabolites (parent:metabolite ratio) in urine and plasma

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Cox-york, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No